CLINICAL TRIAL: NCT00574873
Title: A PHASE 3 RANDOMIZED, OPEN-LABEL STUDY OF BOSUTINIB VERSUS IMATINIB IN SUBJECTS WITH NEWLY DIAGNOSED CHRONIC PHASE PHILADELPHIA CHROMOSOME POSITIVE CHRONIC MYELOGENOUS LEUKEMIA
Brief Title: Compare Bosutinib To Imatinib In Subjects With Newly Diagnosed Chronic Phase Philadelphia Chromosome Positive CML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-3000; B1871008 (Other: Alias Study Number); 2007-003780-50 (EudraCT Number)
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Bosutinib; imatinib; CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bosutinib
  Interventions: Drug: Bosutinib
- 2 (Active Comparator): Imatinib
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: Bosutinib — 500 mg once daily, by mouth (tablet) with food preferably in the morning. Drug can be increased up to 600mg daily in case of lack of efficacy, and can be reduced to 300mg daily in case of toxicity. The drug will be given daily for up to 8 years until treatment failure, unacceptable toxicity, death or withdrawal of consent.
  Other Names: SKI 606
  Arms: 1
Drug: imatinib — 400 mg once daily, by mouth (tablet). Drug can be increased up to 600mg daily in case of lack of efficacy, and can be reduced to 300mg daily in case of toxicity. The drug will be given daily for up to 8 years until treatment failure, unacceptable toxicity, death or withdrawal of consent.
  Other Names: Gleevec
  Arms: 2

SUMMARY:
Two-arm, randomized, open-label trial designed to evaluate the efficacy and safety of bosutinib alone compared to imatinib alone in subjects newly diagnosed with chronic phase Chronic Myelogenous Leukemia (CML). The primary endpoint is cytogenetic response rate at one year.

ELIGIBILITY:
Inclusion Criteria:

* Cytogenetic diagnosis of chronic phase Ph+ CML diagnosed less than 6 months.
* Diagnosis of CML chronic phase confirmed.
* Adequate hepatic and renal function.
* Able to take oral tablets.

Exclusion Criteria:

* Exclusions include Philadelphia negative CML.
* Prior anti-leukemia treatment.
* Prior stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2008-02-05 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2015-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (165):
- United States (32):
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - Tower Cancer Research Foundation (TCRF), Beverly Hills, California
  - Robert A Moss, MD, FACP, Inc, Fountain Valley, California
  - UCSD Medical Center-Thornton, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UCSD Medical Center-Hillcrest, San Diego, California
  - Stanford Hospital and Clinics Investigational Drug Services, Stanford, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Stanford University Medical Center, Stanford, California
  - Cancer Care Centers of Florida, Hudson, Florida
  - Cancer Care Centers of Florida, New Port Richey, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Pasco Pinellas Cancer Center, Tarpon Springs, Florida
  - Northside Hospital, Inc. - GCS/Annex, Atlanta, Georgia
  - Indiana Blood and Marrow Transplantation Research Franciscan St. Francis Health Center Inc., Indianapolis, Indiana
  - Indiana Blood and Marrow Transplantation Research, Indianapolis, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cancer Center of Kansas, Salinas, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Josephine Ford Cancer - Downriver, Brownstown, Michigan
  - Henry Ford Medical Center- Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Hospital - West Bloomfield, Detroit, Michigan
  - Regional Cancer Care Associates, Cherry Hill, New Jersey
  - Study Supplies: Regional Cancer Care Associates, Cherry Hill, New Jersey
  - Somerset Hematology Oncology Associates, Somerville, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Associates In Oncology and Hematology, Chattanooga, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Argentina (4):
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Hospital Privado de Cordoba, Córdoba, Prov. de Cordoba
  - Centro de Investigaciones Oncologicas, Bahía Blanca, Provincia Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
- Belgium (6):
  - Cliniques Universitaires Saint Luc, Brussels
  - C.H.R.ST. - R. Fabiola (N-D), Charleroi
  - University Hospital Gent - Department of Hematology, Ghent
  - Centre Hospitalier de Jolimont - Lobbes, La Louvière
  - CHU de Charleroi - Hopital civil Marie Curie, Lodelinsart
  - H.-Hartziekenhuis Roeselare-Menen, Roeselare
- Centro De Hematologia E Hemoterapia Da Unicamp, Campinas/ SP, Brazil
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
- Chile (2):
  - Instituto Oncologico del Sur, Temuco
  - Instituto Oncologico, Viña del Mar
- China (4):
  - Ruiging Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, P.R. China
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing
  - The Chinese PLA General Hospital, Beijing
  - The Hematology Hospital of Chinese Academy of Medical Science, Tianjin
- Colombia (3):
  - Fundacion Santa Fe de Bogota, Bogota, Cundinamarca
  - Fundacion Cardiovascular de Colombia, Floridablanca, Santander Department
  - CIOSAD Centro de Investigaciones Oncologicas, Bogotá
- France (10):
  - Institut Bergonie, Bordeaux
  - CHU Caen - Cote de Nacre, Caen
  - Centre Hospitalier de Versailles Hopital Andre Mignot, Le Chesnay
  - Hopital EDOUARD HERRIOT, Lyon
  - Hopital HOTEL DIEU, Nantes
  - Hospital Archet 1, Nice
  - Centre d'Investigation Clinique- CIC INSERM802, Poitiers
  - CHU de Poitiers, Poitiers
  - Clinique Sainte Anne, Strasbourg
  - Hopitaux Universitaires de Strasbourg - Hopital Civil, Strasbourg
- Germany (6):
  - Charite University Medical Center - Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Univeristatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig Zentrum fur Innere Medizin, Leipzig
  - III. Medizinische Klinik, Universitaetsklinikum Mannheim gGmbH, Mannheim
  - III. Medizinischen Klinik und Poliklinik des Klinikums Rechts der Isar der TU-MUNCHEN, München
- Prince Of Wales Hospital, Shatin N.T., HONG KONG, Hong Kong
- Hungary (4):
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointezet, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Kaposi Mor Oktato Korhaz, Belgyogyaszati Osztaly, Kaposvár
  - Josa Andras Hospital, Nyíregyháza
- India (5):
  - Tata Memorial Center, Tata Memorial Hospital, Mumbai, Maharashtra
  - Advanced Centre for Treatment, Research and Education in Cancer, Mumbai, Maharashtra
  - Jehangir Clinical Development Centre,, Pune, Maharashtra
  - Birla Cancer Centre, Jaipur, Rajasthan
  - SEAROC Cancer Center, Soni Manipal Hospital, Jaipur, Rajasthan
- Italy (4):
  - Azienda Ospedaliera San Gerardo, Monza, Lombardy
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Ospedale Ferrarotto - Divisione di Ematologia, Catania
  - Dipartimento Di Ematologia Ospedale Santo Eugenio, Roma
- Japan (16):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Tohoku Univesity Hospital, Sendai, Miyagi
  - Kinki University School Of Medicine, Sayama, Osaka
  - Jikei University Hospital Daisan, Komae-shi, Tokyo
  - Japanese Red Cross Nagoya First Hospital, Aichi
  - Aichi Cancer Center Hospital, Aichi
  - Chiba University Hospital, Chiba
  - Tokai University Hospital, Kanagawa
  - Nagasaki University Hospital, Nagasaki
  - Niigata University Medical and Dental Hospital, Niigata
  - Osaka University Hospital, Osaka
  - Hamamatsu Medical University Hospital Faculty of Medicine, Shizuoka
  - Tokyo Metropolitan Cancer & Infectious Disease Centre Komagome Hp, Tokyo
- Riga Centre Of Haematology, Riga, Latvia
- Hematology, Oncology & Transfusion Medicine Center, Vilnius, Lithuania
- Centro Medico de las Americas, Mérida, Mexico
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Im. A. Mieleckiego Slaskiego Uniwersytetu Medycznego, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
- Russia (16):
  - GUZ Komi Republican Oncology Center, Syktyvkar, Komi
  - Regional State Budgetary Healthcare Institution "Barnaul City Hospital #8", Barnaul
  - Kirov Research Institute of Hematology and Blood Transfusion of, Kirov
  - Federal State Budget Institution Hematology Scientific Center of Minzdravsotsrazvitiya of Russia, Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Perm Territory State Budgetary Healthcare Inst, Perm
  - Republican Hospital na Baranov, Petrozavodsk
  - Rostov Regional Clinical Hospital, Rostov-on-Don
  - Rostov State Medical University of the Minzdravsotsrazvitiya of Russia, Rostov-on-Don
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - St-Petersburg Pavlov's State Medical University, Saint Petersburg
  - St-Petersburg State Medical University, Saint Petersburg
  - Samara Regional Clinical Hospital M.I. Kalinin, Samara
  - Yaroslavl Region State Budgetary Healthcare Institution Regional Clinical Hospital, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
  - Central City Hospital #7, Yekaterinburg
- Singapore General Hospital, Singapore, Singapore
- South Africa (5):
  - University Witwatersrand and Oncology, Johannesburg
  - Johannesburg Hospital, Department of Medical Oncology, Parktown
  - Clinical Haematology Unit - Department of Medicine, Soweto
  - Department of Cardiology, Chris Hani Baragwanath Hospital, Soweto
  - Department of Radiology, Chris Hani Baragwanath Hospital, Soweto
- The Catholic University of Korea, Seoul St. Mary's Hospital/Division of Hematology, Seoul, South Korea
- Spain (6):
  - Hospital Universitari Clinic de Barcelona, Barcelona
  - Hospital De La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Madrid Norte-Sanchinarro Centro Integral Oncologico, Madrid
  - Complejo Hospitalario de Toledo- Servicio de Hematologia., Toledo
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
- Taiwan (2):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei TOC
- Division of Hematology, Department of Medicine, Bangkoknoi, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Hacettepe Universitesi Tip Fakultesi, Ankara, Sihhiye
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Gaziantep Universitesi Tip Fakultesi, Gaziantep
- Ukraine (13):
  - Cherkaskiy oblasniy onkologichniy dispanser, Cherkassy
  - Clinical Assocation of Emergency Care, Dnipropetrovsk
  - Clinical Diagnostic Laboratory of Komunalnyj Zaklad, Dnipropetrovsk
  - Komunalnyj Zaklad "Dnipropetrovska Miska Bagatoprofilna Klinichna Likarnja #4", Dnipropetrovsk
  - Instytut Nevidkladnoi ta Vidnovnoi Hirurgii im. P.K. Husaka NAMN Ukrainy, Viddilennja Hematologii, Donetsk
  - Oleksandrovska clinical hospital cardiological rehabilitation department, Kiev
  - Institut Klinichnoi Radiologii DU "Natsionalnyj Naukovyj Centr Radiacijnoi Medicini NAMN Ukraini", Kyiv
  - Institut Klinichnoi Radiologii Naukovogo Centru Radiacijnoi Medicini NAMN Ukraini, Kyiv
  - Institut Klinichnoi Radiologii Naukovogo, Kyiv
  - Miska klinichna likarnja # 9, Kyiv
  - Ultrasaund Educational and Diagnostic Center, Lviv
  - Instutut Patologii Krovi to Transfuziynoi Medicinu AMN Ukraini, Lviv
  - Polyclinic of 5th Municipal Hospital, Lviv
- United Kingdom (8):
  - 3rd Floor Centre for Clinical Haematology, Nottingham, EAST Midlands
  - The Park Hospital, Nottingham, EAST Midlands
  - Hammersmith Hospital Clinical Trial Units, Hammersmith, London
  - Good Hope Hospital, Birmingham, WEST Midlands
  - Birmingham Heartlands Hospital, Birmingham, WEST Midlands
  - Department of Haematology - Level 3, Bexley Wing, Leeds, WEST Yorkshire
  - Department of Haematology, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Garrett M, Knight B, Cortes JE, Deininger MW. Population modeling of bosutinib exposure-response in patients with newly diagnosed chronic phase chronic myeloid leukemia. Cancer Med. 2023 Sep;12(17):17981-17992. doi: 10.1002/cam4.6439. Epub 2023 Aug 8. PMID 37553873
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- [Derived] Gambacorti-Passerini C, Cortes JE, Lipton JH, Dmoszynska A, Wong RS, Rossiev V, Pavlov D, Gogat Marchant K, Duvillie L, Khattry N, Kantarjian HM, Brummendorf TH. Safety of bosutinib versus imatinib in the phase 3 BELA trial in newly diagnosed chronic phase chronic myeloid leukemia. Am J Hematol. 2014 Oct;89(10):947-53. doi: 10.1002/ajh.23788. Epub 2014 Jul 21. PMID 24944159
- [Derived] Hsyu PH, Mould DR, Abbas R, Amantea M. Population pharmacokinetic and pharmacodynamic analysis of bosutinib. Drug Metab Pharmacokinet. 2014;29(6):441-8. doi: 10.2133/dmpk.DMPK-13-RG-126. Epub 2014 Jun 10. PMID 24919837 (Retraction: PMID 30922682 Drug Metab Pharmacokinet. 2019 Apr;34(2):163)
- [Derived] Trask PC, Cella D, Powell C, Reisman A, Whiteley J, Kelly V. Health-related quality of life in chronic myeloid leukemia. Leuk Res. 2013 Jan;37(1):9-13. doi: 10.1016/j.leukres.2012.09.013. Epub 2012 Oct 29. PMID 23116602
- [Derived] Cortes JE, Kim DW, Kantarjian HM, Brummendorf TH, Dyagil I, Griskevicius L, Malhotra H, Powell C, Gogat K, Countouriotis AM, Gambacorti-Passerini C. Bosutinib versus imatinib in newly diagnosed chronic-phase chronic myeloid leukemia: results from the BELA trial. J Clin Oncol. 2012 Oct 1;30(28):3486-92. doi: 10.1200/JCO.2011.38.7522. Epub 2012 Sep 4. PMID 22949154
- [Derived] O'Hare T, Zabriskie MS, Eiring AM, Deininger MW. Pushing the limits of targeted therapy in chronic myeloid leukaemia. Nat Rev Cancer. 2012 Jul 24;12(8):513-26. doi: 10.1038/nrc3317. PMID 22825216
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A4-3000&StudyName=Compare%20Bosutinib%20To%20Imatinib%20In%20Subjects%20With%20Newly%20Diagnosed%20Chronic%20Phase%20Philadelphia%20Chromosome%20Positive%20CML

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib: Bosutinib 500 milligram (mg) tablet orally once daily up to 5 years or until treatment failure, unacceptable toxicity, death, withdrawal of consent. Dose adjustments, if needed, included an escalation to bosutinib 600 mg tablet orally once daily or a reduction to bosutinib 300 mg tablet orally once daily.
- Imatinib: Imatinib 400 mg tablet orally once daily up to 5 years or until treatment failure, unacceptable toxicity, death, withdrawal of consent. Dose adjustments, if needed, included an escalation to imatinib 600 mg tablet orally once daily or a reduction to imatinib 300 mg tablet orally once daily.
Period: Overall Study
Arm/Group | Bosutinib | Imatinib
Started | 250 | 252
Treated | 248 | 251
Completed | 12 | 1
Not Completed | 238 | 251
Not completed — Withdrawal by Subject | 18 | 19
Not completed — Investigator request | 18 | 8
Not completed — Death | 15 | 14
Not completed — Lost to Follow-up | 14 | 5
Not completed — Other | 40 | 4
Not completed — Discontinuation of study by sponsor | 5 | 199
Not completed — Blank, site closed per local regulations | 2 | 2
Not completed — Extension Study | 126 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population - included all participants who were randomized to test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosutinib | Imatinib | Total
Number analyzed (Participants) | 250 | 252 | 502
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (14.39) | 45.6 (14.80) | 46.5 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 117 | 218
  Male | 149 | 135 | 284

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) at Year 1
Description: Cytogenetic Response (CyR) is based on the prevalence of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase on a bone marrow (BM) aspirate. CCyR was achieved when there was 0 percent (%) Ph+ metaphases among cells in a BM sample when at least 20 metaphases from a BM sample were analyzed, or less than (<) 1% breakpoint cluster region Abelson protooncogene (Bcr-Abl) fusion product among cells in a BM sample or peripheral blood sample when at least 200 cells were analyzed.
Time Frame: Year 1 (48 weeks)
Population: Intent-to-treat (ITT) population - included all participants who were randomized to test article.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 250 | 252
Percentage of Participants | 70.0 [64.3 to 75.7] | 68.3 [62.5 to 74.0]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; Test type: Superiority or Other; p = 0.667, Stratified Cochran-Mantel-Haenszel — p-value was based on a Cochran Mantel Haenszel test for general association between treatment and responder stratification by Sokal risk group (low, intermediate, high) and region (1 to 3) as determined at time of randomization

2. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Year 1
Description: Molecular response was assessed using Bcr-Abl transcript levels measured by reverse transcriptase polymerase chain reaction (RT-PCR) from peripheral blood. A MMR was defined as a ratio Bcr-Abl/Abl less than or equal to (≤) 0.1% on the international scale (greater than or equal to [≥] 3 log reduction from standardized baseline in ratio of Bcr-Abl to Abl transcripts) with at least 3000 Abl analyzed.
Time Frame: Year 1 (48 weeks)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 250 | 252
Percentage of Participants | 38.0 [32.0 to 44.0] | 25.4 [20.0 to 30.8]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; Test type: Superiority or Other; p = 0.002, Stratified Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining CCyR at 192 Weeks
Description: The Kaplan-Meier curve was generated based the time from the first date of CCyR until the first date of confirmed loss of CCyR, objectively documented, for responders only. Participants without confirmed loss of CCyR were censored at the last valid cytogenetic assessment.
  CyR is based on the prevalence of Ph+ metaphases among cells in metaphase on a bone marrow sample. CCyR was achieved when there was 0% Ph+ metaphases among cells in a BM sample when at least 20 metaphases from a BM sample were analyzed, or <1% Bcr-Abl fusion product among cells in a BM sample or peripheral blood sample when at least 200 cells were analyzed.
  The medians have not been reached in either arm, as such, the premature estimated hazard ratio is provided. Four years rate was displayed since the majority of participants had first CCyR by Year 1.
Time Frame: 192 weeks
Population: Subgroup of participants from ITT population who had CCyR.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 197 | 204
Percentage of Participants | 92.9 [87.8 to 95.9] | 88.9 [83.2 to 92.7]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.31 to 1.31] — Hazard ratio (95% confidence interval) based on the treatment effect (bosutinib compared with imatinib) in a stratified (by Sokal risk group and region at randomization) Cox model for the hazard of the respective event

4. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining Complete Hematologic Response (CHR) at 192 Weeks
Description: The Kaplan-Meier curve was generated based on the first date of confirmed CHR until the first date of loss of CHR, objectively documented, for responders only. Participants without confirmed loss of response were censored at the last valid hematologic assessment.
  CHR must have been of at least 4 weeks in duration confirmed by 2 assessments at least 4 weeks apart and was defined as follows: white blood cells ≤ institutional upper limit of normal, no peripheral blasts or promyelocytes, myelocytes + metamyelocytes <5% in blood, absolute neutrophil count ≥1.0*10^9/L, platelets ≥100 but <450*10^9/L unless related to therapy, <20% basophils in blood and no extramedually involvement (including hepato- or splenomegaly).
  The medians have not been reached in either arm, as such, the premature estimated hazard ratio is provided. Four years rate was displayed since the majority of participants had first CHR by Year 1.
Time Frame: 192 weeks
Population: Subgroup of participants from ITT population who had CHR.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 219 | 242
Percentage of Participants | 91.6 [86.5 to 94.9] | 86.0 [80.7 to 90.0]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.32 to 1.08] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining Derived MMR at 144 Weeks
Description: The Kaplan-Meier curve was generated based on the first date of MMR until the first date loss of MMR, objectively documented, for responders only. Participants without confirmed loss of response were censored at the last valid molecular assessment.
  Molecular response was assessed using Bcr-Abl transcript levels measured by RT-PCR from peripheral blood. MMR is defined as a ratio Bcr-Abl/Abl ≤0.1% on the international scale (≥3 log reduction from standardized baseline in ratio of Bcr-Abl to Abl transcripts) with at least 3000 Abl analyzed.
  The medians have not been reached in either arm, as such, the premature estimated hazard ratio is provided. Three years rate was displayed since the majority of imatinib participants had first MMR by Year 2.
Time Frame: 144 weeks
Population: Subgroup of participants from ITT population who had MMR.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 168 | 170
Percentage of Participants | 94.7 [89.6 to 97.3] | 98.0 [93.8 to 99.3]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; Test type: Superiority or Other; Hazard Ratio (HR) = 3.25, 95% CI 2-sided [0.90 to 11.72] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Cumulative Incidence of On-Treatment Transformation to Accelerated Phase (AP) or Blast Phase (BP) at 192 Weeks
Description: The cumulative incidence curve was generated based on the time from randomization to the first date of transformation to AP or BP while on study treatment adjusting for the competing risk of treatment discontinuation without transformation, for each participant.
  Criteria for transformation to AP: 15 to 29% blasts; ≥30% blasts + promyelocytes; ≥20% basophils in blood or bone marrow; platelets <100*10^9/L (not related to therapy), in blood. Criteria for transformation to BP: ≥30% blasts in blood or bone marrow and extramedullary involvement other than liver or spleen (example: chloromas).
  Time to transformation was calculated as weeks = ([date of first documented occurrence of the event - date of randomization] + 1)/7. If transformation was not obtained, censoring was at the last hematologic assessment or death (whichever was earliest). Participants who were not treated contributed time = 1 day/7. 95% confidence interval for the cumulative incidence is from Gray's method.
Time Frame: 192 weeks
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 250 | 252
Percentage of Participants | 1.6 [0.6 to 4.3] | 4.4 [2.5 to 7.8]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.13 to 1.29] — The hazard ratio (95% confidence interval) is obtained from a Cox model for cause-specific hazard as a function of the covariate treatment (bosutinib compared with imatinib) with stratification by region and Sokal risk group at randomization

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bosutinib | Imatinib
Serious Adverse Events (participants affected / at risk) | 90/248 | 57/251
Other Adverse Events (participants affected / at risk) | 235/248 | 238/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=248) | Imatinib (N=251)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Neutropenia (Blood and lymphatic system disorders) | 2 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 5 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 2
Generalised oedema (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 1
Bronchitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Infected dermal cyst (Infections and infestations) | 1 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Salmonella bacteraemia (Infections and infestations) | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Dissociative disorder (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pregnancy of partner (Social circumstances) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Glaucoma (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Disease progression (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Allergic hepatitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Dermatitis infected (Infections and infestations) | 1 | 0
Eczema infected (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Intrauterine infection (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Exposure via father (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Hepatitis C antibody positive (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cyst removal (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=248) | Imatinib (N=251)
Thrombocytopenia (Blood and lymphatic system disorders) | 70 | 72
Anaemia (Blood and lymphatic system disorders) | 63 | 58
Neutropenia (Blood and lymphatic system disorders) | 35 | 78
Leukopenia (Blood and lymphatic system disorders) | 24 | 57
Eyelid oedema (Eye disorders) | 3 | 20
Diarrhoea (Gastrointestinal disorders) | 174 | 69
Nausea (Gastrointestinal disorders) | 87 | 93
Vomiting (Gastrointestinal disorders) | 86 | 42
Abdominal pain upper (Gastrointestinal disorders) | 38 | 21
Abdominal pain (Gastrointestinal disorders) | 34 | 19
Dyspepsia (Gastrointestinal disorders) | 22 | 17
Fatigue (General disorders) | 38 | 33
Pyrexia (General disorders) | 44 | 34
Oedema peripheral (General disorders) | 14 | 32
Asthenia (General disorders) | 23 | 23
Oedema (General disorders) | 14 | 16
Upper respiratory tract infection (Infections and infestations) | 33 | 24
Nasopharyngitis (Infections and infestations) | 26 | 28
Alanine aminotransferase increased (Investigations) | 85 | 27
Aspartate aminotransferase increased (Investigations) | 70 | 28
Lipase increased (Investigations) | 47 | 29
Blood creatine phosphokinase increased (Investigations) | 23 | 58
Blood alkaline phosphatase increased (Investigations) | 18 | 11
Blood creatinine increased (Investigations) | 14 | 16
Weight increased (Investigations) | 6 | 24
Gamma-glutamyltransferase increased (Investigations) | 16 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 26 | 55
Decreased appetite (Metabolism and nutrition disorders) | 22 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 22
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 61
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 24
Headache (Nervous system disorders) | 33 | 34
Dizziness (Nervous system disorders) | 23 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 9
Rash (Skin and subcutaneous tissue disorders) | 64 | 49
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 9
Lymphopenia (Blood and lymphatic system disorders) | 8 | 16
Periorbital oedema (Eye disorders) | 4 | 38
Abdominal distension (Gastrointestinal disorders) | 8 | 13
Constipation (Gastrointestinal disorders) | 13 | 12
Face oedema (General disorders) | 5 | 15
Bronchitis (Infections and infestations) | 14 | 14
Influenza (Infections and infestations) | 23 | 11
Pharyngitis (Infections and infestations) | 13 | 4
Toothache (Gastrointestinal disorders) | 13 | 4
Amylase increased (Investigations) | 27 | 16
Haemoglobin decreased (Investigations) | 5 | 14
Weight decreased (Investigations) | 16 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 21
Insomnia (Psychiatric disorders) | 10 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 1
Hypertension (Vascular disorders) | 20 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.